CLINICAL TRIAL: NCT05095597
Title: Umbilical Cord Plasma for Treating Endometrial Pathologies (Thin Endometrium / Asherman's Syndrome/ Endometria Atrophy).
Acronym: hSCU-PRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación IVI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001-FIVI-002-IC; 2020-005717-40 (EudraCT Number)
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Asherman Syndrome; Endometrial Atrophy
Keywords: Endometrial pathology; Platelet-rich plasma; Umbilical cord blood; Regenerative medicine
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Intervention Model Description: Recruitment period:
  * Umbilical cord donors: throughout the study. Although the aim is to recruit the maximum number of umbilical cord samples during the first 10±3 months of the study. 30±15 donors will be recruited.
  * Patients (group A and B): from month 4 of the first year until the end of the study.
  * Expected duration of treatment per patient:
  * Group A (arms 1 and 2): 22±8 days (visit 2 to visit 3).
  * Group B: 22±8 days (visit 2 to visit 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Umbilical cord PRP donors (Other): Women who are going to give birth to a healthy live newborn at the Hospital Universitario y Politécnico La Fe.
  Donors will donate their umbilical cord blood to obtain the hUC-PRP. A total of 30±15 donors will be recruited.
  Interventions: Procedure: Umbilical cord blood collection
- Group B- Asherman with PRP treatment and estrogen therapy (Experimental): Women with thin endometrium/endometrial atrophy and/or Asherman's syndrome with fertility problems and reproductive desires, desires that could be achieved by their participation in the present study. A total of 15 patients will be included; all of them will receive the investigational treatment as well as estrogen therapy.
  Interventions: Procedure: Injection of hUC-PRP by hysteroscopy; Drug: Oestraclin; Procedure: Endometrial biopsy
- Group A1- POI with PRP treatment and estrogen therapy (Other): Women with premature ovarian failure (POI). A total of 10 patients will be included. All of them will receive the investigational treatment as well as estrogen therapy.
  Interventions: Procedure: Injection of hUC-PRP by hysteroscopy; Drug: Oestraclin; Procedure: Endometrial biopsy
- Group A2- POI with estrogen therapy (Other): Women with premature ovarian failure (POI). A total of 10 patients will be included. All of them will receive the estrogen therapy.
  Interventions: Drug: Oestraclin; Procedure: Endometrial biopsy
- Group A3- POI without PRP treatment nor estrogen therapy (Other): Women with premature ovarian failure (POI). A total of 10 patients will be included. None of them will receive either the investigational treatment nor estrogen therapy.
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Injection of hUC-PRP by hysteroscopy — PRP previously frozen at -80ºC (6±2 mL) will be defrozen after checking donor-receptor compatibility and viral safety study. PRP (4±2 mL) will be activated with 5% CaCl2 and immediately injected (4±2 mL) in the sub-endometrial wall via hysteroscopy.
  Arms: Group A1- POI with PRP treatment and estrogen therapy; Group B- Asherman with PRP treatment and estrogen therapy
Drug: Oestraclin — Patients will receive estrogenic therapy, based on estradiol, for 10±2 days (oestraclin, topical cream, 5µg daily for 10±2 days).
  Arms: Group A1- POI with PRP treatment and estrogen therapy; Group A2- POI with estrogen therapy; Group B- Asherman with PRP treatment and estrogen therapy
Procedure: Umbilical cord blood collection — The SCU will be collected using a blood collection bag containing anticoagulant. This step will be performed by the medical and nursing staff of the obstetrics service of the HUP La Fe. The blood collection bags will be the following, or similar: Cord Blood Collection Bags from MACOPHARMA; CPD Umbilical Cord Bag from GRIFOLS.
  Arms: Umbilical cord PRP donors
Procedure: Endometrial biopsy — Biopsies will be taken by specialized medical personnel by aspiration with an intrauterine cannula (pipelle or cornier). Samples will be collected in 15 mL tubes (or in a larger capacity container if needed) containing PBS or RNA later until frozen at -80ºC, at the IVI Foundation facilities. Prior to freezing (in a 1.8-2 mL cryotube) the PBS will be removed and the sample cleaned in a Petri dish if needed.
  Arms: Group A1- POI with PRP treatment and estrogen therapy; Group A2- POI with estrogen therapy; Group A3- POI without PRP treatment nor estrogen therapy; Group B- Asherman with PRP treatment and estrogen therapy

SUMMARY:
In the last years, platelet-rich plasma (PRP) has emerged as a promising alternative to treat endometrial pathologies affecting the endometrial lining. Different studies have tried this therapeutic approach in human patient, but results are not conclusive at all. Also, in the last years, different studies have suggested the umbilical cord blood has a stronger reservoir of growth factors and other pro-regenerative molecules than the adult peripheral blood. That is the reason why the present study aims to evaluate if using platelet-rich plasma obtained from umbilical cord blood is able to increase endometrial thickness and prepare the endometrium for an embryo transference. However, due to the novelty of this approach, the investigators have considered to include a 'proof of concept' group (women with premature ovarian insufficiency) to obtain a deeper understanding of the clinical value of this blood derivative.

DETAILED DESCRIPTION:
Phase II clinical trial, designed as a pilot study, single-center and open-label, which aims to study the efficacy of platelet-rich plasma from umbilical cord after injection into a pathological endometrium (thin endometrium, Asherman's Syndrome, endometrial atrophy).

This treatment will be applied to patients with the aforementioned endometrial pathologies (group B), as well as to patients with premature ovarian failure (group A), which will serve to study its clinical value in greater detail. Plasma samples as well as endometrial biopsies will be analyzed to try to understand what molecular events are triggered in the endometrial tissue after the application of the treatment under study.

ELIGIBILITY:
UMBILICAL CORD DONORS

Donors of umbilical cord blood will be women (and their partners, if applicable) who give birth to a live newborn(s) in the Gynecology and Obstetrics service of HUP La Fe; the same umbilical cord collection criteria will be followed as standardized in HUP La Fe for the donation of this biological product.

GROUP A

Inclusion Criteria:

* Patient information sheet and signed informed consent.
* Female, acting voluntarily, aged between 18 and 48 years at the time of recruitment.
* BMI ≥ 18 kg/m2 and ≤ 35 kg/m2.
* Patients with premature ovarian failure (amenorrhea prior to 40 years of age and FSH > 40 IU/L).

Exclusion Criteria:

* Active genital infection proven at the time of recruitment; chronic endometritis.
* Known endometrial pathology.
* Psychological disorder that may hinder study follow-up.
* Positive results after viral safety analysis (HBsAg, HBcAb, HCV, HIV1, HIV2, syphilis).
* Presenting any syndrome or condition that, from the principal investigator's point of view, could pose a risk to the study or to the patient.
* Any significant clinical anomaly detected during the recruitment process; simultaneous participation in another clinical study that could affect the objectives of the present study or previous participation in this same study.

GROUP B

Inclusion Criteria:

* Information and signed informed consent.
* female, acting voluntarily, aged between 18 and 48 years at the time of recruitment.
* body mass index (BMI): ≥ 18 kg/m2 and ≤ 35 kg/m2.
* Patients undergoing an assisted reproduction cycle.
* Endometrial thickness < 5mm despite estrogen administration for more than 10 days and/or evidence of Asherman's Syndrome.

Exclusion Criteria:

* Active genital infection proven at the time of recruitment; chronic endometritis.
* Known endometrial pathology.
* Psychological disorder that may hinder study follow-up.
* Positive results after viral safety analysis (HBsAg, HBcAb, HCV, HIV1, HIV2, syphilis).
* Presenting any syndrome or condition that, from the principal investigator's point of view, could pose a risk to the study or to the patient.
* Any significant clinical anomaly detected during the recruitment process; simultaneous participation in another clinical study that could affect the objectives of the present study or previous participation in this same study.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Study of endometrial regeneration and/or improvement in patients with endometrial pathologies (thin endometrium/Asherman's syndrome/endometrial atrophy) treated with platelet-rich plasma from the umbilical cord by endometrial thickeness. | An average of 3 months
  Improvement will be studied in form of tissue thickening (mm), comparing endometrial thickness before and after PRP injection

SECONDARY OUTCOMES:
Proof-of-concept in POI patients by improvement endometrial thickeness. | An average of 3 months
  Improvement will be studied in form of tissue thickening (mm), comparing endometrial thickness before and after PRP injection.
Gene and protein level evaluation of the endometrial biopsies collected. | An average of 3 years
  Different molecular and histological assays will be performed with the biopsies from all the groups.
Study of the molecular composition of the different plasma fractions obtained from collected umbilical cord samples. | An average of 3 years
  Different molecular assays will be performed with the blood samples obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Romeu Villaroya, MD., PhD., Principal Investigator — Hospital La Fe; Irene Cervelló Alcaráz, PhD., Study Director — IVI Foundation/ IIS La Fe
Locations (1):
- Hospital la Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication